CLINICAL TRIAL: NCT05586984
Title: A Prospective, Observational Trial of Transvaginal Uterine Suspension With the New Minimally Invasive Uterine Suspension
Brief Title: Transvaginal Sacrospinous Hysteropexy Versus Laparoscopic Uterine Lateral Suspension
Status: Recruiting | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yu Fang Huang, Professor Yu Fang Huang, National Cheng-Kung University Hospital
Other Study IDs: 111-NCKUH-CTC--IIT
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Pelvic Organ Prolapse; Uterine Prolapse
Keywords: Pelvic organ prolapse; Laparoscopic uterine lateral suspension; Transvaginal sacrospinous ligament fixation
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic uterine lateral suspension: Laparoscopic uterine lateral suspension for apical prolapse. Concomitant anterior and posterior colporrhaphy may be performed.
  Interventions: Procedure: Laparoscopic uterine lateral suspension
- Transvaginal sacrospinous fixation: Uterus-preserving transvaginal sacrospinous fixation for apical prolapse. Concomitant anterior and posterior colporrhaphy may be performed.
  Interventions: Procedure: Transvaginal sacrospinous fixation

INTERVENTIONS:
Procedure: Laparoscopic uterine lateral suspension — Laparoscopic uterine lateral suspension done with four trocar sites. Fix a 1.5cm*32cm mesh to uterus at anterior lower segment and bilateral round ligaments by non-absorbable sutures (Surgilon 2-0, Ethicon, Norderstedt, Germany), and to lateral abdominal fascia by non-absorbable sutures (Prolene 1-0, Ethicon, Norderstedt, Germany). Reperitonization done to avoid mesh exposure in peritoneal cavity. Concomitant anterior and posterior colporrhaphy may be performed.
  Groups: Laparoscopic uterine lateral suspension
Procedure: Transvaginal sacrospinous fixation — Transvaginal sacrospinous fixation done by hand suturing uterus to right sacrospinous ligament with non-absorbable suture (Prolene 1-0, Ethicon, Norderstedt, Germany). Concomitant anterior and posterior colporrhaphy may be performed.
  Groups: Transvaginal sacrospinous fixation

SUMMARY:
Transvaginal or transabdominal surgeries are current choices of uterus-preserving surgeries for pelvic organ prolapse.

Laparoscopic lateral uterine suspension, a modified surgical approach of uterine suspension from bilateral abdominal wall fascia, performed with expected safety and simplicity of surgery besides advantages including small wound incision and fast recovery in laparoscopic surgeries. This trial aim to discuss the therapeutic efficacy, long term safety, and adverse events of laparoscopic lateral uterine suspension and compare with the conventional transvaginal sacrospinous ligament fixation with native tissue repair.

DETAILED DESCRIPTION:
Pelvic organ prolapse can be treated either conservatively or surgically. Patients who are unsatisfied with conservative treatment or with severe symptoms often seek for surgical intervention. Transvaginal or transabdominal surgeries are current choices of uterus-preserving surgeries for pelvic organ prolapse. Laparoscopic sacrohysteropexy is the current trend for laparoscopic surgery, with small incisional wound, fast recovery, and low recurrence rate as advantages. However, laparoscopic sacrohysteropexy is often regarded as time consuming and ous sometimes hazard given the complexity of surgical technique and the anatomy of the presacral region. Few cases with severe complications such as vascular injuries, sacral nerve root injuries, and diskitis had been reported with laparoscopic sacrohysteropexy in previous studies.

Laparoscopic lateral uterine suspension, a modified surgical approach of uterine suspension from bilateral abdominal wall fascia, is therefore proposed in our study. The most significant benefits of this novel approach include safety and simplicity of surgery besides advantages including small wound incision and fast recovery in laparoscopic surgeries. This trial aim to discuss the therapeutic efficacy of laparoscopic lateral uterine suspension and compare with the transvaginal sacrospinous ligament fixation with native tissue repair. Other results include safety and adverse events of laparoscopic lateral uterine suspension in long term follow up.

ELIGIBILITY:
Inclusion Criteria:

* older than 21 years old.
* uterine prolapse stage 2 at least, defined by C point distal to -1cm by POP-Q system.
* patients willing to receive a uterine-preserving surgery for pelvic organ prolapse, and is suitable for anesthesia after evaluation.
* patients who had or had not received conservative treatments for pelvic organ prolapse.
* patients able and willing to finish the questionnaire evaluation.

Exclusion Criteria:

* patient who had received a previous hysterectomy, or is planning on concomitant hysterectomy in the surgery for pelvic organ prolapse.
* patient who had received a previous surgery for pelvic organ prolapse.
* patient with history of adverse events following a synthetic mesh.
* patients with chronic or acute pelvic pain.
* patients who had received abdominal or pelvic irradiation.
* patients who cannot receive either surgery due to comorbidity.
* patients pregnant or with future plan of pregnancy.
* patients with vaginal length less than 5cm.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pelvic organ prolapse, predominantly apical prolapse, who had not received a previous surgical correction, and is willing to receive a uterine-preserving surgery for pelvic organ prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 5 years
  Composite outcome of subjective and objective recurrence of uterine prolapse.

SECONDARY OUTCOMES:
Anatomical outcome | 5 years
  Comparison of total vaginal length (TVL), Ba, Bp points defined by POP-Q system.
Functional outcome | 5 years
  Comparison of urination and defecation functions by Pelvic floor disability index-20 (PFDI-20).
Sexual function outcome | 5 years
  Comparison of sexual function by Female Sexual Function Index (FSFI).
Urodynamic outcome | 6 months
  Comparison of post residual urine amount, uroflowmetry, and 1-hour pad test.

OTHER OUTCOMES:
Safety outcome | 5 years
  Surgery-related complications and mesh-related long term complications.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No